CLINICAL TRIAL: NCT03073850
Title: Antithrombotic Treatment in Patients With Effectively Maintained Sinus Rhythm After Atrial Fibrillation Ablation (The ATEMS-AF Study)
Brief Title: Antithrombotic Treatment in Patients With Effectively Maintained Sinus Rhythm After Atrial Fibrillation Ablation
Acronym: ATEMS-AF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Majority of enrolled patients have withdrawn.
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hong Euy Lim, MD, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KUGH12078-001
Record Dates: First submitted 2017-02-02; First posted 2017-03-08 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Aspirin; Clopidogrel; Anticoagulants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Antiplatelet therapy (Experimental): acetylsalicylic acid (ASA) 100mg or clopidogrel 75mg if intolerant to ASA
  Interventions: Drug: Antiplatelet
- Low-dose OAC therapy (Experimental): Edoxaban of 30mg (Reduced dose of 15mg if body weight < 60kg, CCr< 50 ml/min, concomittant use of P-gp)
  Interventions: Drug: Low dose oral anticoagulant
- Standard-dose OAC therapy (Active Comparator): Edoxaban of 60mg (Reduced dose of 30mg if body weight < 60kg, CCr< 50 ml/min, concomittant use of P-gp)
  Interventions: Drug: Standard dose oral anticoagulant

INTERVENTIONS:
Drug: Antiplatelet — ASA or clopidogrel
  Other Names: aspirin 100mg or clopidogrel 75mg
  Arms: Antiplatelet therapy
Drug: Low dose oral anticoagulant — Edoxaban of 30mg
  Other Names: Edoxaban of 30mg
  Arms: Low-dose OAC therapy
Drug: Standard dose oral anticoagulant — Edoxaban of 60mg
  Other Names: Edoxaban of 60mg
  Arms: Standard-dose OAC therapy

SUMMARY:
The purpose of the study is to investigate the best strategy for long-term stroke prevention in patients who have sinus rhythm after a successful catheter ablation for atrial fibrillation (AF) and who are at risk of thromboembolic events (CHA2DS2-VASc score ≥2). The investigators are going to compare antiplatelet therapy to oral anticoagulation (OAC) with different doses of edoxaban (30mg and 60mg).

DETAILED DESCRIPTION:
The investigators hypothesize that the strategy of OAC will be superior to antiplatelet therapy, but low dose edoxaban (30mg) will be non-inferior to standard dose edoxaban (60mg) for reducing the risk of stroke or systemic embolism in patients who underwent successful AF ablation. Although AF ablation is an effective therapy for reducing and/or eliminating the burden of AF, there may continue to be a risk of late recurrence or asymptomatic recurrence of atrial tachyarrhythmias. Until now, the guideline has recommended the continuation of OAC in patients who are at risk of stroke or systemic embolism based on the CHA2DS2-VASc score, even though they have maintained sinus rhythm. The annual rate of stroke, however, is still lower compared to that predicted by the scoring system, because AF ablation reduced the AF burden by 86% and the remaining episodes were significantly shorter in duration (median 6 minutes) than those pre-ablation reported by the previous study. Based on recent studies which demonstrated that both standard-dose and low-dose non-vitamin K OACs (NOAC) performed equally well with regard to the stroke prevention in patients with AF, low dose NOACs may also be sufficient for stroke prevention of briefly lasting AF episodes after successful AF ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients without evidence of any clinically apparent arrhythmia recurrence during at least six months after last catheter ablation of AF.
* Willing and able to provide informed consent

Exclusion Criteria:

* Patients who do not meet all of the above listed inclusion criteria.
* Patients with significant valvular heart disease or mechanical valve.
* Patients with hypertrophic cardiomyopathy.
* Patients with chronic renal impairment with creatinine clearance rate of < 30 mg/dl.
* Patients with contraindication to long-term OAC.
* Patients who had a stroke within one year prior to enrolment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Freedom rate of stroke or systemic embolism during 2 years after successful AF ablation procedure | 2 year
  Check stroke or systemic embolism through neurologic examination or imaging studies

CONTACTS AND LOCATIONS:
Overall Officials: Hong Euy Lim, Dr., Principal Investigator — Korea University Guro Hospital
Locations (4):
- South Korea (4):
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul